CLINICAL TRIAL: NCT02982694
Title: A Phase II Open-label Study With the Anti-PD-L1 Atezolizumab Monoclonal Antibody in Combination With Bevacizumab in Patients With Advanced Chemotherapy Resistant Colorectal Cancer and MSI-like Molecular Signature
Brief Title: Study With Atezolizumab Plus Bevacizumab in Patients With Chemotherapy Resistant, MSI-like, Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The results of the interim analysis showed that the efficacy in the MSS subgroup (MSI like) is inferior to the expected, and this situation is very unlikely to be reversed if the trial is fully completed.
Sponsor: Vall d'Hebron Institute of Oncology (Other)
Collaborators: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VHIO16001 - EORTC 1604; 2016-002001-19 (EudraCT Number)
Record Dates: First submitted 2016-12-01; First posted 2016-12-05 (Estimated); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: MSI; ColoRectal Cancer; Chemotherapy; Resistance, APC
Keywords: MSI; colorectal; chemotherapy; Bevacizumab; Atezolizumab
MeSH Terms: conditions — Colorectal Neoplasms; Activated Protein C Resistance | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atezolizumab and Bevacizumab (Experimental): Atezolizumab will be administered intravenously at 1200 mg on Day 1 every 3 weeks. The dose of bevacizumab in this study is 7.5 mg/kg administered by IV infusion every 3 weeks on Day 1 of each 21 days cycle. Atezolizumab will be administered first, followed by Bevacizumab, with a minimum of 5 minutes between dosing. The interval between cycle infusions must not be < 10 days.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered 1200 mg in 250 ml 0.9% NaCl IV infusion bag, on day 1 of each cycle of 21 days.
  Other Names: TECENTRIQ
Drug: Bevacizumab — Bevacizumab will be administered 7.5 ml/kg (diluted in 0.9% sodium chloride solution) on day 1 of each 21 days cycle.
  Other Names: Avastin

SUMMARY:
The primary objective of this study is to determine the anti-tumor activity, as measured by overall response rate (ORR) of atezolizumab in combination with bevacizumab in patients with chemotherapy resistant CRC and positivity for MSI-like molecular signature. This is an international, open-label single arm (non-randomized), one-stage phase II trial.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be given according to ICH/GCP and national/local regulations.
* Histological or cytological proof of metastatic CRC.
* Disease progression or relapse after at least one line of treatment for advanced CRC with a fluoropyrimidine containing chemotherapy as single agent or in combination (combinations with oxaliplatin, irinotecan, bevacizumab, and cetuximab or panitumumab are allowed).
* Written documentation of positivity for MSI-like gene signature as determined by Agendia test.
* Unresectable disease, with at least one measurable lesion according to RECIST 1.1.
* Age ≥ 18 years.
* WHO performance status of 0-1.
* Ability and capacity to comply with study and follow-up procedures.
* Adequate hematologic and end-organ function, defined by the following laboratory results obtained within 28 calendar days prior to the first study treatment:
* ANC > 1.5 x 109/L (without granulocyte colony-stimulating factor support within 2 weeks prior to Cycle 1, Day 1)
* WBC counts > 2500/μL
* Platelet count > 100,000/ μL (without transfusion within 2 weeks prior to Cycle 1, Day 1)
* Hemoglobin > 9.0 g/dL
* AST, ALT, and alkaline phosphatase < 2.5 x ULN, with the following exceptions:

  * Patients with documented liver metastases: AST and ALT < 5 x ULN
  * Patients with documented liver or bone metastases: alkaline phosphatase < 5 x ULN Bilirubin <1.5 x ULN. Patients with known Gilbert disease who have serum bilirubin level < 3 x ULN may be enrolled.
* PT and PTT <1.5 x ULN, unless on a stable dose of warfarin
* Serum albumin > 2.5 g/dL
* Creatinine clearance > 30 mL/min (Cockcroft-Gault formula or based on 24-hour urine collection)
* Protein < 2+ on dipstick urinalysis or ≤ 1.0 g in a 24-hour urine collection. All patients with ≥2+ protein on dipstick urinalysis at baseline must undergo a 24-hour urine collection for protein.
* Women of child bearing potential (WOCBP) must have a negative serum pregnancy test before registration.
* Patients of childbearing / reproductive potential should use adequate birth control measures, as defined by the investigator, during the study treatment period and for at least 6 months after the last bevacizumab treatment (for women and men) and 5 months after the last atezolizumab treatment (for women). A highly effective method of birth control is defined as those which result in low failure rate (i.e. less than 1% per year) when used consistently and correctly.
* Female subjects who are breast feeding should discontinue nursing before trial registration and until 6 months after the last bevacizumab treatment and 5 months after the last atezolizumab treatment.

Exclusion Criteria:

* Any treatment with investigational drugs (bevacizumab is not considered investigational drug in CRC) within 28 days prior to Cycle 1, Day 1.
* Previous cytotoxic agent within 14 days of planed treatment initiation.
* Active or untreated CNS metastases as determined by computed tomography (CT) or magnetic resonance imaging (MRI)

  * Note: Patients with treated asymptomatic CNS metastases are eligible, provided they meet all of the following criteria:

    * Evaluable or measurable disease outside the CNS
    * No metastases to midbrain, pons, medulla, cerebellum, or within 10 mm of the optic apparatus (optic nerves and chiasm)
    * No history of intracranial or spinal cord haemorrhage
    * No ongoing requirement for dexamethasone as therapy for CNS disease; anticonvulsants at a stable dose are allowed.
    * No evidence of significant vasogenic edema.
    * No stereotactic radiation, whole-brain radiation or neurosurgical resection within 4 weeks prior to Cycle 1, Day 1.
    * Radiographic demonstration of interim stability (i.e., no progression) between the completion of CNS-directed therapy and the screening radiographic study.
    * Screening CNS radiographic study > 4 weeks since completion of radiotherapy or surgical resection and > 2 weeks since discontinuation of corticosteroids.
* Symptomatic lesions amenable to palliative radiotherapy (e.g., bone metastases or metastases causing nerve impingement) should be treated at least 14 days prior to Cycle 1, Day 1.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently).
* Previous (within the last 5 years) or concurrent malignancies, with the exception of those treated with expected curative outcome as cone-biopsied in situ carcinoma of the cervix, basal cell carcinoma of the skin, localized prostate cancer or ductal carcinoma in situ of the breast.
* Life expectancy of < 12 weeks.
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
* Positive test for human immunodeficiency virus (HIV).
* Active hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test prior to randomization) or hepatitis C.

  * Note: Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible.
* Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
* Active tuberculosis.
* Severe infections within 4 weeks prior to Cycle 1, Day 1, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia.
* Signs or symptoms of infection within 2 weeks prior to Cycle 1, Day 1.
* Received therapeutic oral or IV antibiotics within 2 weeks prior to Cycle 1, Day 1.

  * Note: Patients receiving routine antibiotic prophylaxis (e.g., to prevent chronic obstructive pulmonary disease exacerbation or for dental extraction) are eligible.
* Significant cardiovascular or cerebrovascular disease, such as New York Heart Association cardiac disease (Class II or greater), unstable angina, history of stroke, transient ischemic attack, myocardial infarction or cerebrovascular events within the previous 6 months or unstable arrhythmias within the previous 3 months:
* Patients with known coronary artery disease, arrhythmias, congestive heart failure not meeting the above criteria must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate. Baseline evaluation of left ventricular ejection fraction should be considered for all patients, especially in those with cardiac risk factors and/or history of coronary artery disease.
* Patients with known left ventricular ejection fraction <50%.
* Major surgical procedure within 28 days prior to cycle 1, day 1 (or until the surgical wound is fully healed), or planned procedure or surgery during the study.
* Prior allogeneic stem cell or solid organ transplant.
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications.
* Prior treatment with CD137 agonists, anti-CTLA-4, anti-PD-1, or anti-PD-L1 therapeutic antibody or immune-related pathway-targeting agents.
* Current or recent (within 10 calendar days prior to Cycle 1, Day 1) use of dipyridamole, ticlopidine, clopidogrel, or cilostazol.
* Prophylactic or therapeutic use of low molecular-weight heparin (e.g., enoxaparin), direct thrombin inhibitors, or warfarin are permitted, provided, where appropriate anticoagulation indices are stable. Patients should have been on a stable dose (for therapeutic use) for at least two weeks (or until reaching steady state level of the drug) prior to the first study treatment.
* Inadequately controlled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg) (Anti-hypertensive therapy to achieve these parameters is allowable).
* Prior history of hypertensive crisis or hypertensive encephalopathy.
* Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Cycle 1, Day 1.
* Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the bevacizumab or atezolizumab formulation.
* Evidence of bleeding diathesis or clinically significant coagulopathy (in the absence of therapeutic anticoagulation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-11-24 (Actual); Primary Completion 2020-11-27 (Actual); Study Completion 2020-11-27 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | 36 months from first patient in

SECONDARY OUTCOMES:
Immune-related tumor response | 36 months from first patient in
  the measurement that will be used is ir-RECIST (Immune-Related Response Criteria).
Progression Free Survival | 36 months from first patient in
Overall Survival | 36 months from first patient in
Safety and tolerability (adverse event assessment according to CTCAE v 4.0) | 36 months from first patient in

CONTACTS AND LOCATIONS:
Overall Officials: Josep Tabernero Caturla, Prof, Principal Investigator — Vall d'Hebron Institute of Oncology
Locations (7):
- KU Leuven, Leuven, Belgium
- Italy (2):
  - Ospedale Niguarda CA Granda, Milan
  - Second University of Naples, Naples
- The Netherlands Cancer Institute, Amsterdam, Netherlands
- Spain (3):
  - Institut Català d'Oncologia, Barcelona
  - Vall d'Hebron Institute of Oncology, Barcelona
  - Fundación Investigación Clínico de Valencia, Valencia